CLINICAL TRIAL: NCT04929951
Title: The Effect of Micro Fragmented Adipose Tissue (MFAT) on Shoulder Osteoarthritis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Eugene Roh, Clinical Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 59461
Record Dates: First submitted 2021-06-04; First posted 2021-06-18 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Osteoarthritis Shoulder; Shoulder Pain
MeSH Terms: conditions — Shoulder Pain | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: Micro Fragmented Adipose Tissue (MFAT) on Shoulder Osteoarthritis
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MFAT (Micro Fragmented Adipose Tissue) (Experimental): Intra-articular shoulder injection of autologous Micro Fragmented Adipose Tissue harvested from the thigh using tumescent lipoaspiration and processing with minimal manipulation. This harvested tissue will then be injected into the patient's shoulder.
  Interventions: Biological: Micro Fragmented Adipose Tissue
- Conventional Therapy (Active Comparator): Intra-articular injection of corticosteroid (Triamcinolone 40mg)
  Interventions: Biological: Corticosteroid injection

INTERVENTIONS:
Biological: Micro Fragmented Adipose Tissue — Harvesting of Micro Fragmented Adipose Tissue with intra-articular injection
  Other Names: MFAT
  Arms: MFAT (Micro Fragmented Adipose Tissue)
Biological: Corticosteroid injection — Sham harvesting of adipose tissue without intra-articular injection. Intra-articular injection of corticosteroid.
  Arms: Conventional Therapy

SUMMARY:
This is a non-surgical trial comparing the clinical and functional outcomes of patients with osteoarthritis treated with Intra-articular injection of Micro Fragmented Adipose Tissue versus conventional therapy of intra-articular injection of corticosteroid.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial to compare outcomes between intra-articular injection of Micro Fragmented Adipose Tissue and intra-articular injection of corticosteroid in patients with mild to moderate osteoarthritis of the shoulder. Micro Fragmented Adipose Tissue will be harvested at the subcutaneous tissue by lipoaspiration. Once fat tissue is obtained, it will be processed with minimal manipulation in the clinic room.

To be considered for participation in this study, patients must have radiographic evidence of mild to moderate osteoarthritis of the shoulder (glenohumeral joint). In addition, patients must meet several inclusion/exclusion criteria to be randomized and included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 25 and 75 years-old
* Diagnosis of pre-existing osteoarthritis of the glenohumeral joint
* Working understanding of the English language and able to fully understand the procedure
* Capable of providing informed consent
* Able to complete online, in-person or phone surveys for the purposes of follow-up
* Capable of understanding pre- and post-procedure care instructions
* Ambulatory at baseline
* Previous trial and failure of conservative therapy consisting of a minimum of 6 weeks of physical therapy and trial of anti-inflammatory medications if not contraindicated, with or without concomitant bracing and/or injections.

Exclusion Criteria:

* Age < 25 or > 75 years old
* Radiographs demonstrating either no, little osteoarthritis, severe(bone on bone) osteoarthritis
* Prior total or partial joint replacement surgery or surgery involving cartilage regeneration
* Previous cortisone, PRP or Hyaluronic acid intra-articular injection within the last 3 months
* Co-morbidity with the rheumatologic condition, inflammatory arthritis
* Currently undergoing immunomodulatory therapy
* Uncontrolled endocrine disorder
* BMI >40 or joint space not visible by ultrasound
* Current diagnosis of osteomyelitis, human immunodeficiency virus (HIV-1, -2) and/or hepatitis C (HCV), infection, and poorly controlled diabetes (HgA1C >7.0)
* Pregnancy or planned pregnancy
* previous stem cell injection into treatment joint
* Patient scheduled to undergo any concomitant shoulder surgical procedures or other surgery which may affect outcomes.
* Coagulopathy or anticoagulant treatment
* Chronic pain involving multiple body parts or opioid medication management
* Diagnosis of fibromyalgia
* Concomitant massive(2 tendons with retraction), complete rotator cuff tendon tear

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-07-28 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
ASES Shoulder Score | 24 Months
  Patient reported outcome measure that reports shoulder pain and shoulder functionality

SECONDARY OUTCOMES:
DASH Outcome Measure | 24 Months
  Patient reported questionnaire that measures physical function and symptoms
Veterans RAND 12 (VR-12) score | 24 Months
  Patient reported quality of life outcome measure on a scale of 0-50 with 50 being healthy

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States